CLINICAL TRIAL: NCT02842658
Title: Aerobic Interval Exercise Preconditioning to Prevent Cardiometabolic and Neuropsychological Complications of Anthracycline Based Breast Cancer Chemotherapy
Brief Title: Exercise Preconditioning and Breast Cancer Cardiotoxicity
Acronym: EXACCT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Collaborators: Arizona State University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 15-004656
Record Dates: First submitted 2016-04-15; First posted 2016-07-25 (Estimated); Last update posted 2020-02-24 (Actual); Status verified 2020-02

CONDITIONS: Breast Cancer
Keywords: Chemotherapy; Exercise
MeSH Terms: conditions — Breast Neoplasms; Motor Activity

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- A high-intensity interval exercise group (Active Comparator): Supervised exercise training with be carried out at the Mayo Clinic Cardiac rehabilitation center on cycle ergometers using EKG telemetry. Treatment will begin one week prior to chemotherapy and is tailored around 8 weeks.
  Interventions: Other: A high-intensity interval exercise group
- An attention-control group (Other): Patients will receive counseling regarding physical activity during chemotherapy. Patients will receive a weekly phone call to maintain physical activity during chemotherapy and compliance will be verified using physical activity diaries and pedometers.
  Interventions: Other: An Attention-Control Group

INTERVENTIONS:
Other: A high-intensity interval exercise group — To avoid or reduce muscle soreness or cramps, adequate warm-up is suggested
  Arms: A high-intensity interval exercise group
Other: An Attention-Control Group — Patients will be contacted weekly to access physical activity. To avoid or reduce muscle soreness or cramps, adequate warm-up is suggested
  Arms: An attention-control group

SUMMARY:
The purpose of this study is to determine whether a supervised exercise-training program, initiated prior to chemotherapy induction (pre-conditioning) and continued throughout chemotherapy treatment, can preserve short- and long-term cardiovascular performance, skeletal muscle function, cognitive ability and quality of life better than current standard or care recommendations for exercise during chemotherapy.

DETAILED DESCRIPTION:
The primary aim of this study is to determine the efficacy of a novel, high-intensity aerobic interval exercise preconditioning protocol to ameliorate anthracycline-mediated cardiac and skeletal muscle toxicity in women with breast cancer undergoing de novo chemotherapy.

Research Design:

Women with breast cancer scheduled to undergo de novo chemotherapy with anthracyclines will be enrolled. Qualified patients will be randomized to either 1) a high-intensity interval exercise group, or 2) an attention-control group.

Supervised exercise training will be carried out at the Mayo Clinic Cardiac rehabilitation center in Arizona on cycle ergometers using Electrocardiogram (EKG) telemetry. Patients in the high-intensity interval exercise group will perform four, 4-min intervals at 85-90% peak heart rate (PHR), separated by 3 min at 50% PHR. Each training session will begin with a 10-minute warm-up at 50% of PHR and end with a 5-min cool down at 50% PHR.

The attention-controls will receive counseling consistent with standard of care regarding physical activity during chemotherapy. Attention-control group will receive a weekly phone call to maintain physical activity during chemotherapy and compliance will be verified using physical activity diaries and pedometers.

Treatment for each group will commence 1-week prior to chemotherapy induction. The first dose of chemotherapy will be given within 16-18 hours of the last bout of exercise. High-intensity intermittent exercise (HIIE) training will be continued throughout four, 2-week cycles of chemotherapy (total training time = 9 weeks, 3 days/week).

ELIGIBILITY:
Inclusion Criteria:

* Subjects must be able to communicate meaningfully with the investigator and must be legally competent to provide written informed consent
* Subjects will have been recently diagnosed with breast cancer (stage I, II or III)
* Subjects must be scheduled by their oncologist to undergo anthracycline based chemotherapy (doxorubicin and cyclophosphamide) in the neoadjuvant/adjuvant setting

Exclusion Criteria:

* Unstable angina
* Myocardial infarction in the past 4 weeks
* Uncompensated heart failure
* New York Heart Association class IV symptoms
* Complex ventricular arrhythmias
* Medical orthopedic conditions precluding stationary cycling
* Medical conditions precluding neuropsychological assessment
* Symptomatic severe aortic stenosis
* Acute pulmonary embolus
* Acute myocarditis
* Untreated high-risk proliferative retinopathy
* Recent retinal hemorrhage
* Uncontrolled hypertension
* Sodium and/or Potassium ≥ Grade 2
* Pregnant Women

Ages: 40 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2016-04; Primary Completion 2019-10-18 (Actual); Study Completion 2019-10-18 (Actual)

PRIMARY OUTCOMES:
Change in left ventricular ejection fraction | baseline, approximately 2 months
  Echocardiography will be used to assess biventricular systolic function.
Change in diastolic function | baseline, approximately 2 months
  Echocardiography will be used to assess biventricular diastolic function.

CONTACTS AND LOCATIONS:
Overall Officials: Farouk Mookadam, MBBCh, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Arizona, Scottsdale, Arizona, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials